CLINICAL TRIAL: NCT04895696
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-Controlled, Study to Evaluate the Efficacy and Safety of Afimetoran in Participants With Active Systemic Lupus Erythematosus
Brief Title: A Study Evaluating the Efficacy and Safety of Afimetoran Compared With Placebo in Participants With Active Systemic Lupus Erythematosus (SLE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM026-024; 2023-504320-25-00 (Registry Identifier: EU Trial Number); U1111-1241-6528 (Registry Identifier: UTN)
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: BMS-986256; Systemic Lupus Erythematosus; SLE; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases; Afimetoran
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Afimetoran: Dose 1 (Experimental)
  Interventions: Drug: Afimetoran
- Afimetoran: Dose 2 (Experimental)
  Interventions: Drug: Afimetoran
- Afimetoran: Dose 3 (Experimental)
  Interventions: Drug: Afimetoran
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Afimetoran — Specified dose on specified days
  Other Names: BMS-986256
  Arms: Afimetoran: Dose 1; Afimetoran: Dose 2; Afimetoran: Dose 3
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety and tolerability of Afimetoran in participants with active Systemic Lupus Erythematosus (SLE). The extension period will provide additional long-term safety and efficacy data and enable those participants initially randomized to placebo to receive treatment with Afimetoran.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed ≥ 12 weeks before the screening visit and qualify as having SLE according to the SLE International Collaborating Clinics (SLICC) Classification Criteria at the screening visit
* Test positive, as determined by the central laboratory, for at least one of the following lupus related autoantibodies at the time of screening: antinuclear antibody ≥ 1:80, anti-double-stranded deoxyribonucleic acid (dsDNA) antibody, or anti-Smith antibody.
* Have a total Hybrid Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score ≥ 6 points and clinical Hybrid SLEDAI score ≥ 4 points with joint involvement and/or rash

Exclusion Criteria:

* Active severe lupus nephritis (LN) as assessed by the investigator
* Active or unstable neuropsychiatric lupus manifestations defined by the Hybrid SLEDAI
* Diagnosis of Mixed Connective Tissue Disease for which the predominant diagnosis is not SLE
* Antiphospholipid Syndrome

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2029-04-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants that achieve an SLE (Systemic Lupus Erythematosus) Responder Index (4) (SRI(4)) response at Week 48 | Up to 48 Weeks

SECONDARY OUTCOMES:
Proportion of participants that achieve a British Isles Lupus Assessment Group (BILAG)-based Combine Lupus Assessment (BICLA) response at Week 24 and Week 48 | Up to 48 Weeks
Proportion of participants who achieve an SRI(4) response at Week 24 | Up to 24 Weeks
Proportion of participants who achieve a Lupus Low Disease Activity State (LLDAS) response at Week 24 and Week 48 | Up to 48 Weeks
Proportion of participants with a Cutaneous Lupus Erythematosus Disease Area and Severity Index; Activity (CLASI-A) score ≥ 10 at baseline who achieve a decrease of ≥ 50% from baseline CLASI-A score (CLASI-50) response at Week 24 and Week 48 | Up to 48 Weeks
Proportion of participants with 6 or more swollen joints and 6 or more tender joints at baseline who achieve a ≥ 50% reduction from baseline in both swollen and tender joints at Week 24 and Week 48 | Up to 48 Weeks
Mean change from baseline in swollen joint count using the 28-joint count at Week 24 and Week 48 in participants with ≥ 2 swollen joints at baseline | Up to 48 Weeks
Mean change from baseline in tender joint count at Week 24 and Week 48 using the 28- joint count in participants with ≥ 2 tender joints at baseline | Up to 48 Weeks
Change from baseline in PGA score of disease activity at Week 24 and Week 48 | Up to 48 Weeks
  PGA = Physician Global Assessment of disease activity (score of "0" indicating no disease activity and higher scores indicating higher disease activity)
Proportion of participants who achieve CS reduction or maintenance to ≤ 7.5 mg per day at Week 48 | Up to 48 Weeks
Change in participant reported disease activity from baseline to Week 24 and Week 48 according to the 36-item Short Form Health Questionnaire (SF-36) | Up to 48 Weeks
  The SF-36 was designed as an indicator of health status in population surveys, and health policy evaluations, and for use as an outcome measure in clinical practice and research. Scores for each domain range from 0 to 100, with high scores indicating a better health status.
Number of participants with Adverse Events (AEs) | Up to 100 Weeks
Number of participants with Serious Adverse Events (SAEs) | Up to 100 Weeks
Number of participants with clinical laboratory abnormalities | Up to 100 Weeks
Number of participants with physical examination abnormalities | Up to 100 Weeks
Number of participants with vital sign abnormalities | Up to 100 Weeks
Number of participants with electrocardiogram (ECG) abnormalities | Up to 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (147):
- United States (36):
  - Local Institution - 0100, Birmingham, Alabama
  - Local Institution - 0123, Huntington Beach, California
  - Local Institution - 0170, La Jolla, California
  - Local Institution - 0159, La Palma, California
  - Local Institution - 0172, San Diego, California
  - Local Institution - 0164, Woodland Hills, California
  - Local Institution - 0121, Clearwater, Florida
  - Local Institution - 0167, Kissimmee, Florida
  - Local Institution - 0122, Orlando, Florida
  - Local Institution - 0173, Ormond Beach, Florida
  - Local Institution - 0154, Plantation, Florida
  - Local Institution - 0137, South Miami, Florida
  - Local Institution - 0155, Tamarac, Florida
  - Local Institution - 0160, Atlanta, Georgia
  - Local Institution - 0205, Suwanee, Georgia
  - Local Institution - 0146, Orland Park, Illinois
  - Local Institution - 0187, Hopkinsville, Kentucky
  - Local Institution - 0171, Baton Rouge, Louisiana
  - Local Institution - 0134, Wheaton, Maryland
  - Local Institution - 0070, Eagan, Minnesota
  - Local Institution - 0124, St Louis, Missouri
  - Local Institution - 0165, St Louis, Missouri
  - Local Institution - 0091, Las Vegas, Nevada
  - Local Institution - 0219, West Long Branch, New Jersey
  - Local Institution - 0140, Manhasset, New York
  - Local Institution - 0132, The Bronx, New York
  - Local Institution - 0203, Charlotte, North Carolina
  - Local Institution - 0103, Charlotte, North Carolina
  - Local Institution - 0151, Columbus, Ohio
  - Local Institution - 0042, Middleburg Heights, Ohio
  - Local Institution - 0152, Allen, Texas
  - Local Institution - 0197, Allen, Texas
  - Local Institution - 0136, Amarillo, Texas
  - Local Institution - 0029, Mesquite, Texas
  - Local Institution - 0163, San Antonio, Texas
  - Local Institution - 0223, Bellevue, Washington
- Argentina (9):
  - Local Institution - 0130, Quilmes, Buenos Aires
  - Local Institution - 0195, San Fernando, Buenos Aires
  - Local Institution - 0025, Córdoba, Córdoba Province
  - Local Institution - 0074, Buenos Aires, Distrito Federal
  - Local Institution - 0040, CABA, Distrito Federal
  - Local Institution - 0027, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0207, Buenos Aires
  - Local Institution - 0128, Buenos Aires
  - Local Institution - 0041, San Juan
- Australia (6):
  - Local Institution - 0063, Botany, New South Wales
  - Local Institution - 0072, Westmead, New South Wales
  - Local Institution - 0066, Maroochydore, Queensland
  - Local Institution - 0065, Woodville, South Australia
  - Local Institution - 0062, Camberwell, Victoria
  - Local Institution - 0064, Ivanhoe, Victoria
- Brazil (9):
  - Local Institution - 0006, Salvador, Estado de Bahia
  - Local Institution - 0031, Salvador, Estado de Bahia
  - Local Institution - 0093, Cuiabá, Mato Grosso
  - Local Institution - 0008, Juiz de Fora, Minas Gerais
  - Local Institution - 0010, Curitiba, Paraná
  - Local Institution - 0007, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0014, São Bernardo do Campo, São Paulo
  - Local Institution - 0045, São José do Rio Preto, São Paulo
  - Local Institution - 0009, São Paulo
- Chile (5):
  - Local Institution - 0127, Osorno, Los Lagos Region
  - Local Institution - 0143, Valdivia, Los Ríos Region
  - Local Institution - 0075, Providencia, Santiago Metropolitan
  - Local Institution - 0073, Santiago, Santiago Metropolitan
  - Local Institution - 0043, Santiago, Santiago Metropolitan
- China (10):
  - Local Institution - 0177, Beijing, Beijing Municipality
  - Local Institution - 0180, Beijing, Beijing Municipality
  - Local Institution - 0184, Shenzhen, Guangdong
  - Local Institution - 0176, Nanjing, Jiangsu
  - Local Institution - 0188, Nanjing, Jiangsu
  - Local Institution - 0193, Suzhou, Jiangsu
  - Local Institution - 0174, Changchun, Jilin
  - Local Institution - 0179, Dalian, Liaoning
  - Local Institution - 0178, Jinan, Shandong
  - Local Institution - 0183, Jining, Shandong
- Colombia (6):
  - Local Institution - 0190, Medellín, Antioquia
  - Local Institution - 0001, Barranquilla
  - Local Institution - 0004, Bogotá
  - Local Institution - 0076, Cali
  - Local Institution - 0005, Chía
  - Local Institution - 0003, Zipaquirá
- France (7):
  - Local Institution - 0156, Pessac, Aquitaine
  - Local Institution - 0083, Brest, Finistère
  - Local Institution - 0048, Bordeaux
  - Local Institution - 0144, Caen
  - Local Institution - 0129, Lille
  - Local Institution - 0112, Marseille
  - Local Institution - 0044, Strasbourg
- Germany (4):
  - Local Institution - 0087, Cologne, North Rhine-Westphalia
  - Local Institution - 0085, Berlin
  - Local Institution - 0086, Essen
  - Local Institution - 0084, Freiburg im Breisgau
- India (5):
  - Local Institution - 0226, Ahmedabad, Gujarat
  - Local Institution - 0214, Gurugram, Haryana
  - Local Institution - 0210, Bengaluru, Karnataka
  - Local Institution - 0208, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0209, Secunderabad, Telangana
- Ireland (3):
  - Local Institution - 0119, Manorhamilton, Leitrim
  - Local Institution - 0106, Dublin
  - Local Institution - 0107, Galway
- Japan (16):
  - Local Institution - 0114, Eiheiji-cho,Yoshida-gun, Fukui
  - Local Institution - 0095, Kitakyushu, Fukuoka
  - Local Institution - 0096, Sapporo, Hokkaido
  - Local Institution - 0104, Kanazawa, Ishikawa-ken
  - Local Institution - 0099, Sendai, Miyagi
  - Local Institution - 0117, Bunkyo-ku, Tokyo
  - Local Institution - 0218, Fuchū, Tokyo
  - Local Institution - 0113, Itabashiku, Tokyo
  - Local Institution - 0150, Meguro-ku, Tokyo
  - Local Institution - 0098, Shinjuku-ku, Tokyo
  - Local Institution - 0105, Shinjuku-ku, Tokyo
  - Local Institution - 0138, Aichi
  - Local Institution - 0115, Chiba
  - Local Institution - 0162, Fukushima
  - Local Institution - 0097, Tokyo
  - Local Institution - 0116, Tokyo
- Mexico (9):
  - Local Institution - 0020, León, Guanajuato
  - Local Institution - 0017, Guadalajara, Jalisco
  - Local Institution - 0022, Zapopan, Jalisco
  - Local Institution - 0060, Mexico City, Mexico City
  - Local Institution - 0018, Mexico City, Mexico City
  - Local Institution - 0071, Monterrey, Nuevo León
  - Local Institution - 0021, Chihuahua City
  - Local Institution - 0158, Mexico City
  - Local Institution - 0061, Mérida
- Poland (4):
  - Local Institution - 0204, Warsaw, Masovian Voivodeship
  - Local Institution - 0049, Poznan
  - Local Institution - 0149, Warsaw
  - Local Institution - 0052, Wroclaw
- Local Institution - 0037, San Juan, Puerto Rico
- Romania (4):
  - Local Institution - 0082, Râmnicu Vâlcea, Vâlcea County
  - Local Institution - 0157, Bucharest
  - Local Institution - 0067, Bucharest
  - Local Institution - 0068, Giroc
- Spain (5):
  - Local Institution - 0206, Santander, Cantabria
  - Local Institution - 0056, A Coruña
  - Local Institution - 0058, Barcelona
  - Local Institution - 0055, Madrid
  - Local Institution - 0057, Seville
- Taiwan (5):
  - Local Institution - 0080, Kaohsiung Niao Sung Dist
  - Local Institution - 0081, Taichung
  - Local Institution - 0078, Taichung
  - Local Institution - 0079, Taipei
  - Local Institution - 0077, Taipei
- United Kingdom (3):
  - Local Institution - 0111, Cambridge, Cambridgeshire
  - Local Institution - 0110, Bradford
  - Local Institution - 0125, Manchester

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04895696.html